CLINICAL TRIAL: NCT02327052
Title: Assessment of Speckle Tracking Strain Predictive Value for Myocardial Fibrosis in Subjects With Chagas Disease
Brief Title: Assessment of Speckle Tracking Strain Predictive Value for Myocardial Fibrosis in Chagas Disease
Status: Completed | Type: Observational
Sponsor: Hospital Sao Rafael (Other)
Responsible Party: Principal Investigator, Milena Botelho Pereira Soares, Assessment of Speckle Tracking Strain Predictive Value for Myocardial Fibrosis in Subjects with Chagas Disease, Hospital Sao Rafael
Other Study IDs: PCL01-04
Record Dates: First submitted 2014-12-18; First posted 2014-12-30 (Estimated); Results first posted 2021-03-24 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Chagas Disease
Keywords: Chagas disease; longitudinal global strain; speckle tracking
MeSH Terms: conditions — Chagas Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Chagas disease: The study comprised 58 subjects with Chagas disease, confirmed by two positive serologic tests.
  Interventions: Other: No intervention was performed.

INTERVENTIONS:
Other: No intervention was performed. — No intervention was performed.

SUMMARY:
One of the most challenging issues of chronic Chagas disease is to provide earlier detection of heart involvement. Two-dimensional speckle tracking (2-D ST) echocardiography, a new imaging modality with useful applications in several cardiac diseases, has been validated for subjects with myocardial infarction against cardiac magnetic resonance (CMR). Here the investigators hypothesize that the longitudinal global strain (LGS) has an incremental value to ejection fraction for predicting myocardial fibrosis in subjects with Chagas disease.

DETAILED DESCRIPTION:
We conducted a cross-sectional study, in which adult subjects with Chagas disease were invited to participate. From January 2011 to December 2013, we included 58 subjects from a convenience sample, in the Chagas disease outpatient clinics at our institution. Inclusion criteria were disease established based on microbiological confirmation by two positive serologic tests (indirect hemagglutination and indirect immunofluorescence), and age between 18 and 70 years. Exclusion criteria were: previous myocardial infarction or history of coronary artery disease; primary valve disease; dialysis treatment of terminal renal failure, liver disease in activity; hematologic, neoplastic or bone diseases; and MRI contraindications.

The study complied with the Declaration of Helsinki and was approved by the Ethics Committee of the Hospital São Rafael. All subjects gave written informed consent before their inclusion in the study.

We obtained a structured medical history, and all subjects underwent physical examination, blood analysis, 12-lead ECG, chest X-Ray, 24-h Holter monitoring, conventional Doppler echocardiogram plus speckle tracking strain, and cardiac magnetic resonance.

Doppler echocardiogram Standard transthoracic echocardiographic examinations were recorded in all subjects using the Vivid 7 digital ultrasound system (GE Vingmed Ultrasound AS, Horten, Norway). Three cardiac cycles were stored in cine loop format for online analysis. LV and left atrial dimensions were measured according to the American Society of Echocardiography's recommendations [13]. The LV EF was measured using the biplane Simpson's method. S0 systolic velocity at the lateral mitral annulus was assessed using pulsed-wave DTI. Diastolic function was evaluated by the analysis of the mitral Doppler inflow, pulsed- wave DTI at the lateral mitral annulus, and mitral propagation velocity using color M-mode echocardiography. Mitral regurgitation (MR) was obtained using the proximal isovelocity surface area method. Right ventricular function was assessed with the S0 systolic velocity in the lateral wall. Systolic pulmonary arterial pressure was obtained from the tricuspid regurgitation flow. In subjects with adequate Doppler MR signals, dP/dt was determined noninvasively from the rate of change of MR velocity, according to American Society of Echocardiography guidelines.

Strain Measurements Two-dimensional gray-scale images were acquired in the standard apical four-chamber, three-chamber, and two-chamber views at a frame rate of 80 frames/sec. The dimensions of the computation area were an angle of 80o and at a depth of 13 cm. The left ventricle was divided into 17 segments, and each segment was analyzed individually. GLS and segmental longitudinal strain were obtained as previously described [14]. Average longitudinal strains were calculated automatically by the software. Two-dimensional strain is a non-Doppler-based method for the evaluation of systolic strain using standard 2D acquisitions. After placing three endocardial markers in an end-diastolic frame, the software automatically tracks the contour on subsequent frames. Adequate tracking can be verified in real time and corrected by adjusting the region of interest or by manually correcting the contour to ensure optimal tracking. Two-dimensional longitudinal strain was assessed in apical views. Average longitudinal strains were calculated for the 17 segments.

Magnetic resonance imaging Cardiac magnetic resonance exams were performed on all subjects using the General Electric Sigma HDx 1.5-T system (Fairfield, CT, USA). Images were acquired and gated to the ECG during breath-hold, four-chamber, short axis and long axis of the left ventricle, in the exact same location in different sequences. This allows a precise comparison between cardiac function and regional myocardial structure. The parameters used in the dynamic sequences were repetition time (RT) of 3.5 ms, echo time (ET) of 1.5 ms, flip angle 60°, bandwidth of receipt of ± 125 kHz, field of view (FOV) of 35 x 35 cm, 256x148 matrix, temporal resolution (TR) 35 ms, 8.0 mm slice thickness, without a space between the slices. Following this acquisition, a dose of gadolinium-based contrast (0.1 mmol / kg) was injected. The myocardial delayed enhancement (MDE) technique was used to investigate myocardial fibrosis, an inversion-recovery pre-pared gradient-echo acquired 10 to 20 min after contrast application, with the following parameters: Repetition time (RT) 7.1 ms, echo time (ET) 3.1 ms, flip angle 20°, cardiac phases 1, views per segment 16 to 32, matrix 256 X 192, slice thickness 8 mm, gap between slices 2 mm and field of view 32 to 38 cm, inversion time 150 to 300 ms, receiver bandwidth 31.25 kHz, number of excitations 2, acquisition every heart beat. The mass of fibrosis was estimated by a quantitative visual method.

Statistical analysis Categorical data were presented as numbers (percentages), and continuous data were expressed as mean (SD) or median (interquartile range). Comparisons of continuous variables among groups were performed with analysis of variance (ANOVA) test or Kruskal-Wallis, depending on normality assessed by Shapiro-Wilk test. Chi-Square or Fisher tests were applied for proportions comparisons. Correlations between continuous variables were evaluated by Pearson or Spearman coefficients, depending on normality. Receiver-operating characteristic (ROC) curve analysis was used to evaluate if the longitudinal global strain would add accuracy to the ejection fraction in the predicted fibrosis. C-Statistic (area under the curve) was presented as a unified estimate of sensitivity and specificity. To determine the ability to predict myocardial fibrosis, multiple linear regression was performed, adjusting longitudinal global strain to left ventricular ejection fraction. Analyses in subgroups with normal and low ejection fraction were also accomplished. Cases with missing data were not included in the analysis. Analyses were performed using SPSS version 20.0 (IBM), and p < 0.05 (two-tailed) was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Chagas disease, established based on microbiological confirmation by two positive serologic tests (indirect hemagglutination and indirect immunofluorescence)
* Between 18 and 70 years of age.

Exclusion Criteria:

* Previous myocardial infarction or history of coronary artery disease
* Primary valve disease
* Dialysis treatment of terminal renal failure
* Liver disease in activity
* Hematologic, neoplastic or bone diseases
* And MRI contraindications.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult subjects in the Chagas disease outpatient clinics at our institution from January 2011 to December 2013 were invited to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2011-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Milena Soares, PhD, Principal Investigator — Hospital São Rafael
Locations (1):
- Hospital São Rafael, Salvador, Estado de Bahia, Brazil

RESULTS

PARTICIPANT FLOW:
Groups:
- Chagas Disease: The study comprised 58 subjects with Chagas disease, confirmed by two positive serologic tests, from a convenience sample.
Period: Overall Study
Arm/Group | Chagas Disease
Started | 58
Completed | 58
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Chagas Disease: See below Baseline Measures
Arm/Group | Chagas Disease
Number analyzed (Participants) | 58
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 58
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 24
Region of Enrollment [Number; unit: participants]
  Brazil | 58

OUTCOME MEASURES:

1. Primary Outcome: Correlation Between Longitudinal Global Strain and the Percentage of Myocardial Fibrosis on Magnetic Resonance
Description: Longitudinal global strain were assesseb by standard transthoracic echocardiographic examinations were recorded in all subjects using the Vivid 7 digital ultrasound system (GE Vingmed Ultrasound AS, Horten, Norway) and myocardial fibrosis by cardiac magnetic resonance exams were performed on all subjects using the General Electric Sigma HDx 1.5-T system (Fairfield, CT, USA).
  .
Time Frame: Both outcome measures will be assessed at one month of follow up.
Measure: Mean (Standard Deviation); unit: percentage of fibrosis
Arm/Group | Chagas Disease
Number analyzed (Participants) | 58
percentage of fibrosis | 16.8 (5.5)

ADVERSE EVENTS:
Time Frame: No intervention was performed and we conducted a cross-sectional study, therefore adverse events were not monitored
Description: No intervention was performed and we conducted a cross-sectional study, therefore adverse events were not monitored
Groups:
- Chagas Disease: No intervention was performed and we conducted a cross-sectional study, therefore there were no adverse events.
Arm/Group | Chagas Disease
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No